CLINICAL TRIAL: NCT03519581
Title: Micropulse for Suppression of Diabetic Macular Edema
Acronym: PULSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: IRIDEX Corporation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1141752
Record Dates: First submitted 2018-04-26; First posted 2018-05-09 (Actual); Results first posted 2024-12-17 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Diabetic Macular Edema
Keywords: DME; micropulse laser

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Subjects will be masked to their treatment assignment. The research coordinator that performs the measurement of best corrected visual acuity will be masked to the treatment assignment. The reading center analyst responsible for reviewing and analyzing OCT and microperimetry reports will be masked to treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Micropulse Laser Treatment (Active Comparator): Subjects assigned to the micropulse laser arm of the trial will undergo the following procedures:
  1. Confirmation of the subject's identity and eye to be treated
  2. Subject's eye will be dilated
  3. Subject will be positioned at the slit lamp for treatment
  4. Application of subthreshold micropulse laser using the Iridex IQ577 laser unit. (intermittent pulsed energy) in a 7 X 7 grid pattern surrounding the fovea.
  Interventions: Device: Micropulse Laser Treatment
- Sham Treatment (Placebo Comparator): Subjects assigned to the sham arm of the trial will undergo the following procedures:
  1. Confirmation of the subject's identity and eye to be treated
  2. Subject's eye will be dilated
  3. Subject will be positioned at the slit lamp for treatment
  4. No Actual laser treatment will occur
  Interventions: Device: Sham Treatment

INTERVENTIONS:
Device: Micropulse Laser Treatment — Participant's study eye will be dilated prior to being comfortably seated at the slit lamp for treatment. Application of micropulse laser on retinal surface will occur using TxCell Scanning Delivery System in a 7 x 7 grid to surround the fovea.
  Arms: Micropulse Laser Treatment
Device: Sham Treatment — Participant's study eye will be dilated prior to being comfortably seated at the slit lamp for treatment. No actual laser treatment will occur.
  Arms: Sham Treatment

SUMMARY:
Diabetic retinopathy is one of the most common complications of diabetes and diabetic macular edema (DME) is one of the most common causes of vision loss in diabetes.

The purpose of this study is to determine if early intervention with micropulse laser treatment in eyes with good visual acuity (20/32 or better) will improve or stabilize vision loss due to the complications of diabetic macular edema.

DETAILED DESCRIPTION:
This is a randomized, controlled clinical trial comparing subthreshold micropulse laser versus sham laser treatment for eyes with diabetic macular edema with good visual acuity of 20/32 or better.

Subjects will be randomized to receive either subthreshold micropulse laser treatment or no treatment (sham). Randomization will occur as a ratio of 2:1 and will take place during the clinic visit.

Subjects selected for the study will undergo a complete ophthalmic examination, including measurements of best corrected visual acuity, low luminance visual acuity, contrast sensitivity (using ETDRS testing with a masked coordinator), intraocular pressure, slit lamp exam including documentation of lens status, and dilated funduscopic exam with standard dilating agents used at the UC Davis Eye Center. Subjects will then undergo baseline imaging including Spectral Domain Ocular Coherence Tomography (SD-OCT), fundus autofluorescence (FAF) and microperimetry testing. Both the use of OCT, FAF, and microperimetry testing are within the standard of care for the management of DME.

The duration of an individual subject's participation in the study will be two years which will include at least 10 total visits at various time points including on the day of enrollment, followed by 1, 3, 6, 9, and 12, 15, 18, 21, 24 months after the day of enrollment.

The subjects in the treatment arm will be treated on the day of randomization by SML photocoagulation using the Iridex IQ577 laser unit with TxCell scanning laser delivery system.

Subjects in the sham treatment arm will undergo the same set up procedures as those receiving the laser treatment, however, no actual laser treatment will occur.

Subjects will then return to the clinic for repeat ophthalmic exam, OCT imaging, and microperimetry at 1 month, 3 month, 6 month, 9 month, 12 month, 15 month, 18 month, 21 month and 24 month time points, which is similar in frequency as standard of care.

Patients in the treatment arm are eligible for repeat SML laser at any subsequent visit if there is any decline in vision (1 or more ETDRS lines) or worsening in edema (>10% increase), at the discretion of the treating physician. If vision declines to 20/40 or worse at any study visit, patients in the treatment arm will undergo repeat treatment with SML laser, while those in the sham arm will undergo repeat sham laser.

ELIGIBILITY:
Inclusion Criteria:

1. Age >=18 years
2. Type 1 or type 2 diabetes mellitus
3. Clinical evidence of center-involved DME confirmed on OCT, and defined by OCT

   Central Subfield (CSF) thickness at the time of randomization by the following:
   1. Zeiss Cirrus: 275μ in women, and 290μ in men
   2. Heidelberg Spectralis: 290μ in women, and 305μ in men
4. Best corrected visual acuity of 20/32 or better on ETDRS testing

Exclusion Criteria:

1. Macular edema from causes other than DME
2. An ocular condition is present such that in the opinion of the investigator, visual acuity would not improve from resolution of macular edema (i.e/foveal atrophy, pigment abnormalities, dense hard exudates)
3. An ocular condition is present other than DME which may contribute to macular edema (i.e/vein occlusion, ERM, uveitis, RP, etc…).
4. Cataract that in the opinion of the investigator may alter visual acuity throughout the course of the study
5. History of prior laser or other surgical, intravitreal, or peribulbar treatment for DME in the study eye within the prior 6 months.
6. More than 4 prior intraocular injections for treatment of DME at any time
7. More than 1 prior focal/grid macular photocoagulation session for treatment of DME at any time
8. History of topical steroid or NSAID treatment within 30 days prior to randomization
9. History of PRP within 4 months prior to randomization or anticipated need for PRP in the 6 months following randomization.
10. Any history of vitrectomy.
11. History of major ocular surgery (cataract extraction, scleral buckle, any intraocular surgery, etc.) within prior 4 months or anticipated within the next 6 months following randomization
12. History of YAG capsulotomy performed within 2 months prior to randomization.
13. Aphakia
14. Exam evidence of external ocular infection, including conjunctivitis, chalazion, or significant blepharitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-04-20 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Yiu, MD, PhD, Principal Investigator — University of California, Davis
Locations (1):
- University of California, Davis, Sacramento, California, United States

REFERENCES:
- See also: Learn more or sign up for the study here! — https://studypages.com/s/a-study-of-experimental-treatment-with-micropulse-for-diabetic-macular-edema-build-up-of-fluid-in-the-eye-317967/

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Eyes
Groups:
- Micropulse Laser Treatment: Eyes assigned to the micropulse laser arm of the trial will undergo the following procedures:
  1. Confirmation of the subject's identity and eye to be treated
  2. Subject's eye will be dilated
  3. Subject will be positioned at the slit lamp for treatment
  4. Application of subthreshold micropulse laser using the Iridex IQ577 laser unit. (intermittent pulsed energy) in a 7 X 7 grid pattern surrounding the fovea.
  Micropulse Laser Treatment: Participant's study eye will be dilated prior to being comfortably seated at the slit lamp for treatment. Application of micropulse laser on retinal surface will occur using TxCell Scanning Delivery System in a 7 x 7 grid to surround the fovea.
- Sham Treatment: Eyes assigned to the sham arm of the trial will undergo the following procedures:
  1. Confirmation of the subject's identity and eye to be treated
  2. Subject's eye will be dilated
  3. Subject will be positioned at the slit lamp for treatment
  4. No Actual laser treatment will occur
  Sham Treatment: Participant's study eye will be dilated prior to being comfortably seated at the slit lamp for treatment. No actual laser treatment will occur.
Period: Overall Study
Arm/Group | Micropulse Laser Treatment | Sham Treatment
Started | 16; 16 Eyes (19 total participants enrolled (27 eyes). Some participants had 1 eye enrolled in treatment and the other eye enrolled in sham, therefore the number showing in the "total participants" is not accurate.) | 11; 11 Eyes (19 total participants enrolled (27 eyes). Some participants had 1 eye enrolled in treatment and the other eye enrolled in sham, therefore the number showing in the "total participants" is not accurate.)
Completed | 2; 2 Eyes | 2; 2 Eyes
Not Completed | 14; 14 Eyes | 9; 9 Eyes
Not completed — Lost to Follow-up | 3 | 2
Not completed — Adverse Event | 5 | 2
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Change to insurance | 2 | 1
Not completed — Other | 2 | 4

BASELINE CHARACTERISTICS:
Population: Sex: male, female
Units Other Than Participants: Eyes
Groups:
- Micropulse Laser Treatment: Subjects assigned to the micropulse laser arm of the trial will undergo the following procedures:
  1. Confirmation of the subject's identity and eye to be treated
  2. Subject's eye will be dilated
  3. Subject will be positioned at the slit lamp for treatment
  4. Application of subthreshold micropulse laser using the Iridex IQ577 laser unit. (intermittent pulsed energy) in a 7 X 7 grid pattern surrounding the fovea.
  Micropulse Laser Treatment: Participant's study eye will be dilated prior to being comfortably seated at the slit lamp for treatment. Application of micropulse laser on retinal surface will occur using TxCell Scanning Delivery System in a 7 x 7 grid to surround the fovea.
- Sham Treatment: Subjects assigned to the sham arm of the trial will undergo the following procedures:
  1. Confirmation of the subject's identity and eye to be treated
  2. Subject's eye will be dilated
  3. Subject will be positioned at the slit lamp for treatment
  4. No Actual laser treatment will occur
  Sham Treatment: Participant's study eye will be dilated prior to being comfortably seated at the slit lamp for treatment. No actual laser treatment will occur.
- Total: Total of all reporting groups
Arm/Group | Micropulse Laser Treatment | Sham Treatment | Total
Number analyzed (Participants) | 16 | 11 | 19
Number analyzed (Eyes) | 16 | 11 | 27
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: 19 participants were enrolled. Of those 19 participants, 11 had only one eye enrolled. This accounts for the row population difference.
  Years | 57.1 (8.4) | 54.9 (10.9) | 56.2 (9.3)
Sex: Female, Male [Count of Units; unit: Eyes]
  Female | 6 | 4 | 10
  Male | 10 | 7 | 17
Race (NIH/OMB) [Count of Units; unit: Eyes]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 8 | 4 | 12
  White | 8 | 6 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Best Corrected Visual Acuity (BCVA) [Mean (Standard Deviation); unit: ETDRS Letters Read] | 81.8 (5.0) | 82.5 (4.0) | 82.1 (4.5)
Low Luminance Visual Acuity (LLVA) [Mean (Standard Deviation); unit: EDTDRS Letters Read] | 38.8 (7.5) | 40.6 (7.61) | 39.5 (7.5)
Contrast Sensitivity (CS) [Mean (Standard Deviation); unit: unit less] — The contrast sensitivity chart (CS) uses letters whose contrast varies from high to low. The scale is 0.0 (minimum) to 2.0 (maximum). A higher score equates to a better outcome. The score is based on the contrast of the last group in which 2 or 3 letters were correctly read. A score of 2.0 indicates normal CS of 100%. Scores < than 2.0 signify poorer CS; scores < than 1.5 is consistent with visual impairment; a score < than 1.0 represents visual disability.
  unit less | 1.58 (0.16) | 1.61 (0.17) | 1.59 (0.16)
Central Subfield Thickness (CST) [Mean (Standard Deviation); unit: microns] | 329.7 (23.9) | 354.9 (76.6) | 340.0 (52.4)
Microperimetry Average Threshold [Mean (Standard Deviation); unit: decibels (dB)] | 24.8 (1.9) | 24.5 (2.1) | 24.6 (2.0)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Vision Loss to 20/40 or Worse
Description: BCVA measured using ETDRS testing. The study endpoint was reached if the study patient experienced vision loss of ≥10 letters (≥2 lines) at any visit or 5-9 letters (1-2 lines) at 2 consecutive visits ≤28 days apart, based on the criteria for initiating anti-VEGF therapy as defined in the DRCR Protocol V study.
Time Frame: 6 months
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Micropulse Laser Treatment | Sham Treatment
Number analyzed (Participants) | 16 | 11
Number analyzed (Eyes) | 16 | 11
Eyes | 5 | 3
Statistical Analysis 1: Comparison: Micropulse Laser Treatment vs Sham Treatment; The target sample size for the study was 30 eyes, based on power calculations to achieve 80% power assuming 40% of sham-treated eyes will reach the vision loss threshold within 2 years, while SML treatment will reduce that value to 15%, using a 2:1 ratio for randomization (2 treatment : 1 sham); Test type: Other — The primary statistical analysis was an intention-to-treat analysis. The primary outcome was analyzed by Kruskal-Wallis test because the data was non-parametric; p = .76, Kruskal-Wallis

2. Secondary Outcome: Visual Acuity at 6 Month
Description: Visual acuity measured using ETDRS
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Letters Read
Units Other Than Participants: Eyes
Arm/Group | Micropulse Laser Treatment | Sham Treatment
Number analyzed (Participants) | 16 | 11
Number analyzed (Eyes) | 16 | 11
Letters Read | 79.4 (8.0) | 83.9 (6.3)
Statistical Analysis 1: Comparison: Micropulse Laser Treatment vs Sham Treatment; Test type: Superiority; p = .16, t-test, 2 sided

3. Secondary Outcome: Low Luminance Visual Acuity at 6 Months
Description: Low Luminance Visual acuity measured with a 2.0-log unit neutral density filter
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Letters Read
Units Other Than Participants: Eyes
Arm/Group | Micropulse Laser Treatment | Sham Treatment
Number analyzed (Participants) | 16 | 11
Number analyzed (Eyes) | 16 | 11
Letters Read | 30.7 (13.5) | 40.1 (5.4)
Statistical Analysis 1: Comparison: Micropulse Laser Treatment vs Sham Treatment; Test type: Superiority; p = .12, t-test, 2 sided

4. Secondary Outcome: Contrast Sensitivity at 6 Months
Description: Contrast sensitivity is measured using a single, large letter size (20/60 optotype) with contrast varying across groups of letters. The contrast sensitivity chart (CS) uses letters whose contrast varies from high to low. The scale is 0.0 (minimum) to 2.0 (maximum). A higher score equates to a better outcome. The score is based on the contrast of the last group in which 2 or 3 letters were correctly read. A score of 2.0 indicates normal CS of 100%. Scores < than 2.0 signify poorer CS; scores < than 1.5 is consistent with visual impairment; a score < than 1.0 represents visual disability.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: unit less
Units Other Than Participants: Eyes
Arm/Group | Micropulse Laser Treatment | Sham Treatment
Number analyzed (Participants) | 16 | 11
Number analyzed (Eyes) | 16 | 11
unit less | 1.54 (.21) | 1.61 (.23)
Statistical Analysis 1: Comparison: Micropulse Laser Treatment vs Sham Treatment; Test type: Superiority; p = .68, t-test, 2 sided

5. Secondary Outcome: Central Subfield Thickness (CST) at 6 Months
Description: Using Heidelberg Spectralis device to measure central subfield thickness (CST)
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: microns
Units Other Than Participants: Eyes
Arm/Group | Micropulse Laser Treatment | Sham Treatment
Number analyzed (Participants) | 16 | 11
Number analyzed (Eyes) | 16 | 11
microns | 357.8 (90.4) | 356.9 (50.0)
Statistical Analysis 1: Comparison: Micropulse Laser Treatment vs Sham Treatment; Test type: Superiority; p = .96, t-test, 2 sided

6. Secondary Outcome: Microperimetry Average Threshold at 6 Month
Description: Performed using the Macular Integrity Assessment (MAIA) Instrument
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: dB
Units Other Than Participants: Eyes
Arm/Group | Micropulse Laser Treatment | Sham Treatment
Number analyzed (Participants) | 16 | 11
Number analyzed (Eyes) | 16 | 11
dB | 22.5 (3.9) | 24.4 (3.9)
Statistical Analysis 1: Comparison: Micropulse Laser Treatment vs Sham Treatment; Test type: Superiority — Two-tailed t-tests and mixed effects regression models; p = .50, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Micropulse Laser Treatment | Sham Treatment
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/11
Other Adverse Events (participants affected / at risk) | 5/16 | 2/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Micropulse Laser Treatment (N=16) | Sham Treatment (N=11)
Worsening Diabetic Macular Edema (Eye disorders) | 2 (2) | 0 (0)
Vitreous Hemorrhage (Eye disorders) | 1 (1) | 1 (1)
Posterior Vitreous Detachment (Eye disorders) | 1 (1) | 0 (0)
Decrease in Visual Acuity (Eye disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-10-06): https://cdn.clinicaltrials.gov/large-docs/81/NCT03519581/Prot_002.pdf
  • Informed Consent Form (2021-03-10): https://cdn.clinicaltrials.gov/large-docs/81/NCT03519581/ICF_001.pdf